CLINICAL TRIAL: NCT03650387
Title: Open-label, Multicenter, Uncontrolled, Rater-blinded, Post-market Clinical Follow-up [PMCF] Study to Confirm Performance and Safety of RADIESSE® (+) Lidocaine in the Treatment of Nasolabial Folds, Marionette Lines, and/or Cheek Volume Loss
Brief Title: Safety, Effectiveness and Participant Satisfaction Study of a Dermal Filler (of RADIESSE® (+) Lidocaine) in the Treatment of Ageing Signs in the Face
Acronym: RaLido
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Collaborators: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M900391005
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Signs of Facial Aging With Volume Loss in the Upper Cheeks, Nasolabial Folds and Marionette Lines

STUDY DESIGN:
Masking Description: Rater-blinded live evaluation of scale scores (the blinded rater does not know which indications were treated)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- RADIESSE® (+) Lidocaine (Experimental)
  Interventions: Device: RADIESSE® (+) Lidocaine

INTERVENTIONS:
Device: RADIESSE® (+) Lidocaine — RADIESSE® (+) Lidocaine will be injected as per its current approved labelling and investigator's usual practice
  Other Names: Radiesse® Injectable Dermal Filler with Lidocaine

SUMMARY:
The primary objective is to collect clinical data to confirm performance and safety for RADIESSE® (+) Lidocaine, when used in accordance with its labelling in the treatment of nasolabial folds, marionette lines and/or upper cheek volume loss.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female greater than or equal to (>=) 18 years old.
2. Participants seeking for dermal filler/volumising treatment in at least two of the following indications:

   * Nasolabial folds;
   * Marionette lines;
   * Cheek volume loss.
3. Nasolabial folds volume deficit of moderate to very severe intensity (grade 2 to 4) on the Merz Nasolabial Folds Scale with symmetrical rating at Day 1 as determined by the blinded rater and confirmed by the treating investigator afterwards.
4. Marionette lines volume deficit of moderate to very severe intensity (grade 2 to 4) on the Merz Marionette Lines Scale with symmetrical rating at Day 1 as determined by the blinded rater and confirmed by the treating investigator afterwards.
5. Upper cheek volume deficit of moderate to very severe intensity (grade 2 to 4) on the Merz Upper Cheek Fullness Scale with symmetrical rating at Day 1 as determined by the blinded rater and confirmed by the treating investigator afterwards.

At least two of the inclusion criteria 3, 4, and 5 must be fulfilled. Depending on the fulfilled criteria, the respective indications will be treated.

Exclusion Criteria:

1. Any prior treatment with silicone, polymethyl methacrylate, fat injections, poly L-lactic acid or permanent dermal fillers in the face.
2. Any prior facial surgery, including facial plastic surgery, thread lift, any unknown treatment, or any surgical permanent implant that could interfere with performance assessments.
3. Prior treatment within the past 24 months with porcine based collagen fillers or with volumisers (e.g., Belotero® Volume or others) in the area to be treated.
4. Prior treatment within the past 18 months with calcium hydroxylapatite in the area to be treated.
5. Prior treatment within the past 12 months with hyaluronic acid in the area to be treated.
6. Prior treatment within the past 6 months with facial dermal therapies (e.g. epilation, ultraviolet irradiation, radiofrequency, facial ablative or non-ablative laser treatment, microderm abrasion, mechanical or chemical peels, non-invasive skin-tightening [e.g., Ultherapy, Thermage] or surgical procedures) or plans to receive this during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (7):
- Germany (7):
  - Rosenpark Research, Merz Investigational Site #490099, Darmstadt
  - Universität Hamburg Fachbereich Chemie Institut für Biologie und Molekularbiologie , Merz Investigational Site #490095, Hamburg
  - Derma Science GmbH Hamburg, Merz Investigational Site #490345, Hamburg
  - Privatpraxis für Dermatologie und Ästhetik, Merz Investigational Site #490371, Munich
  - Dermatologie München-Neuhausen, Merz Investigational Site #490372, Munich
  - Haut-und Lasercentrum, Merz Investigational Site #0490362, Potsdam
  - Centroderm GmbH, Merz Investigational Site #490367, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pavicic T, Sattler G, Fischer T, Dirschka T, Kerscher M, Gauglitz G, Dersch H, Kravtsov M, Heide I, Prager W. Calcium Hydroxyapatite Filler With Integral Lidocaine CaHA (+) for Soft Tissue Augmentation: Results from an Open-Label Multicenter Clinical Study. J Drugs Dermatol. 2022 May 1;21(5):481-487. doi: 10.36849/JDD.6737. PMID 35533030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The multicenter study was conducted at 7 investigational sites in Germany.
Pre-assignment Details: A total of 209 participants were screened, out of which 207 participants were enrolled and treated.
Groups:
- RADIESSE® (+) Lidocaine: All Participants: Participants received study medical device (SMD) (RADIESSE® [+] Lidocaine) on Day 1 with volume for each area to be treated and using injection techniques based on investigator's judgement, skin conditions, safety and participant's expectations. A minimum of two and a maximum of three indications (nasolabial folds, marionette lines, cheek volume loss) per participant were treated. An optional touch-up was performed at Week 4 (Visit 2) in the indications that were treated on Day 1, to obtain an optimal aesthetic outcome, as appropriate.
Period: Overall Study
Arm/Group | RADIESSE® (+) Lidocaine: All Participants
Started | 207
Completed | 173
Not Completed | 34
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 12
Not completed — Adverse Event (Not related) | 1
Not completed — Due to COVID-19 Pandemic | 8

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) was the subset of all participants who were exposed to the SMD at least once.
Groups:
- RADIESSE® (+) Lidocaine: All Participants: Participants received SMD (RADIESSE® [+] Lidocaine) on Day 1 with volume for each area to be treated and using injection techniques based on investigator's judgement, skin conditions, safety and participant's expectations. A minimum of two and a maximum of three indications (nasolabial folds, marionette lines, cheek volume loss) per participant were treated. An optional touch-up was performed at Week 4 (Visit 2) in the indications that were treated on Day 1, to obtain an optimal aesthetic outcome, as appropriate.
Arm/Group | RADIESSE® (+) Lidocaine: All Participants
Number analyzed (Participants) | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (10.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 205
  Asian | 0
  Black or African American | 2
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate for Nasolabial Folds Based on the Blinded Rater's Evaluation on the Merz Nasolabial Folds Scale (MNLFS) at Week 12/16 (Depending on Touch-up)
Description: The MNLFS was used to assess the severity of nasolabial folds. The assessment was performed separately for the left and the right nasolabial fold by the blinded rater and the treating investigator (at baseline only prior to SMD injection) by live rating. MNLFS was a 5 point scale ranging as: 0 (no folds), 1 (mild folds), 2 (moderate folds), 3 (severe folds), 4 (very severe folds). Responders rate was defined as percentage of participants who achieved improvement of greater than or equal to (>=) 1 point in both folds (left and right) from Day 1 pre-injection to Week 12/16 (depending on touch-up). As planned, the cumulative data was collected for Week 12 or Week 16 based on the touch-up.
Time Frame: At Week 12 (for participants with no touch-up) or Week 16 (for participants with touch-up)
Population: The full analysis set (FAS) was the subset of all participants who were exposed to the SMD at least once and for whom a baseline and a post-baseline Merz Aesthetics Scales (MAS) value of at least one treated indication was available. This outcome measure (OM) was analyzed only for participants treated for nasolabial folds.
Measure: Number; unit: percentage of participants
Groups:
- RADIESSE® (+) Lidocaine: Nasolabial Folds: Participants received SMD (RADIESSE® [+] Lidocaine) on Day 1 with volume and using injection techniques based on investigator's judgement, skin conditions, safety and participant's expectations, and the extent of the volume loss/deficit for treatment of nasolabial folds. An optional touch-up was performed at Week 4 (Visit 2) in the indications that were treated on Day 1, to obtain an optimal aesthetic outcome, as appropriate.
Arm/Group | RADIESSE® (+) Lidocaine: Nasolabial Folds
Number analyzed (Participants) | 202
percentage of participants | 93.6
Statistical Analysis 1: Comparison: RADIESSE® (+) Lidocaine: Nasolabial Folds; Test type: Other; p < 0.0001, Exact one-sample binomial test — Bonferroni-Holm was used for alpha correction; The one-sample binomial test was used to test whether the probability of being a responder (p) is significantly above 60%

2. Primary Outcome: Responder Rate for Marionette Lines Based on the Blinded Rater's Evaluation on the Merz Marionette Lines Scale (MMLS) at Week 12/16 (Depending on Touch-up)
Description: The MMLS was used to assess the severity of marionette lines. The assessment was performed separately for the left and the right marionette line by the blinded rater and the treating investigator (at baseline only prior to SMD injection) by live rating. MMLS was a 5 point scale ranging as: 0 (no lines), 1 (mild lines), 2 (moderate lines), 3 (severe lines), 4 (very severe lines). Responders rate was defined as percentage of participants who achieved improvement of >=1 point in both marionette lines (left and right) from Day 1 pre-injection to Week 12/16 (depending on touch-up). As planned, the cumulative data was collected for Week 12 or Week 16 based on the touch-up.
Time Frame: At Week 12 (for participants with no touch-up) or Week 16 (for participants with touch-up)
Population: The FAS was the subset of all participants who were exposed to the SMD at least once and for whom a baseline and a post-baseline MAS value of at least one treated indication was available. This OM was analyzed only for participants treated for marionette lines.
Measure: Number; unit: percentage of participants
Groups:
- RADIESSE® (+) Lidocaine: Marionette Lines: Participants received SMD (RADIESSE® [+] Lidocaine) on Day 1 with volume and using injection techniques based on investigator's judgement, skin conditions, safety and participant's expectations, and the extent of the volume loss/deficit for treatment of marionette lines. An optional touch-up was performed at Week 4 (Visit 2) in the indications that were treated on Day 1, to obtain an optimal aesthetic outcome, as appropriate.
Arm/Group | RADIESSE® (+) Lidocaine: Marionette Lines
Number analyzed (Participants) | 194
percentage of participants | 88.7
Statistical Analysis 1: Comparison: RADIESSE® (+) Lidocaine: Marionette Lines; Test type: Other; p < 0.0001, Exact one-sample binomial test — Bonferroni-Holm was used for alpha correction; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Responder Rate for Cheek Fullness Based on the Blinded Rater's Evaluation on the Merz Upper Cheek Fullness Scale (MUCFS) at Week 12/16 (Depending on Touch-up)
Description: The MUCFS was used to assess the severity of volume loss of upper cheeks. The assessment was performed separately for the left and the right cheek by the blinded rater and the treating investigator (at baseline only prior to SMD injection) by live rating. MUCFS was a 5 point scale ranging as: 0 (full upper cheek), 1 (mildly sunken upper cheek), 2 (moderately sunken upper cheek), 3 (severely sunken upper cheek), 4 (very severely sunken upper cheek). Responders rate was defined as percentage of participants who achieved improvement of >=1 point in both cheeks (left and right) from Day 1 pre-injection to Week 12/16 (depending on touch-up). As planned, the cumulative data was collected for Week 12 or Week 16 based on the touch-up.
Time Frame: At Week 12 (for participants with no touch-up) or Week 16 (for participants with touch-up)
Population: The FAS was the subset of all participants who were exposed to the SMD at least once and for whom a baseline and a post-baseline MAS value of at least one treated indication was available. This OM was analyzed only for participants treated for cheek volume loss.
Measure: Number; unit: percentage of participants
Groups:
- RADIESSE® (+) Lidocaine: Cheek Volume Loss: Participants received SMD (RADIESSE® [+] Lidocaine) on Day 1 with volume and using injection techniques based on investigator's judgement, skin conditions, safety and participant's expectations, and the extent of the volume loss/deficit for treatment of upper cheek volume loss. An optional touch-up was performed at Week 4 (Visit 2) in the indications that were treated on Day 1, to obtain an optimal aesthetic outcome, as appropriate.
Arm/Group | RADIESSE® (+) Lidocaine: Cheek Volume Loss
Number analyzed (Participants) | 188
percentage of participants | 81.9
Statistical Analysis 1: Comparison: RADIESSE® (+) Lidocaine: Cheek Volume Loss; Test type: Other; p < 0.0001, Exact one-sample binomial test — Bonferroni-Holm was used for alpha correction; [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: Number of Participants Reporting One or More Treatment Emergent Adverse Events (TEAEs)
Time Frame: Baseline up to Week 72 (for participants with no touch-up) or Week 76 (for participants with touch-up)
Population: The SES was the subset of all participants who were exposed to the SMD at least once. This OM was analyzed in all participants and by the subpopulations of each indication (participants treated for nasolabial folds, for marionette lines, and for cheek volume loss).
Measure: Count of Participants; unit: Participants
Groups:
- RADIESSE® (+) Lidocaine: All Participants: Participants received SMD (RADIESSE® [+] Lidocaine) on Day 1 with volume and using injection techniques based on investigator's judgement, skin conditions, safety and participant's expectations and depended on the area to be treated for minimum of two and a maximum of three indications (nasolabial folds, marionette lines, cheek volume loss). An optional touch-up was performed at Week 4 (Visit 2) in the indications that were treated on Day 1, to obtain an optimal aesthetic outcome, as appropriate. Participants were included in multiple reporting arms as per treated indications. All participants reporting arm represented all treated participants.
Arm/Group | RADIESSE® (+) Lidocaine: Nasolabial Folds | RADIESSE® (+) Lidocaine: Marionette Lines | RADIESSE® (+) Lidocaine: Cheek Volume Loss | RADIESSE® (+) Lidocaine: All Participants
Number analyzed (Participants) | 203 | 195 | 189 | 207
Participants | 139 | 133 | 129 | 142

5. Secondary Outcome: Responder Rate for Nasolabial Folds Based on the Blinded Rater's Evaluation on the MNLFS at Week 4 (Prior to Optional Touch-up), at Week 24/28, at Week 48/52, and at Week 72/76 (Depending on Touch-up)
Description: The MNLFS was used to assess the severity of nasolabial folds. The assessment was performed separately for the left and the right nasolabial fold by the blinded rater and the treating investigator (at baseline only prior to SMD injection) by live rating. MNLFS was a 5 point scale ranging as: 0 (no folds), 1 (mild folds), 2 (moderate folds), 3 (severe folds), 4 (very severe folds). Responders rate was defined as percentage of participants who achieved improvement of >=1 point in both folds (left and right) from Day 1 pre-injection to Week 4, Week 24/28, Week 48/52, and Week 72/76 (depending on touch-up). As planned, the cumulative data was collected for Week 24 or 28, Week 48 or 52, and Week 72 or 76 based on the touch-up.
Time Frame: At Week 4 (prior to optional touch-up); at Weeks 24, 48 and 72 (for participants with no touch-up) or at Weeks 28, 52 and 76 (for participants with touch-up)
Population: The FAS was the subset of all participants who were exposed to the SMD at least once and for whom a baseline and a post-baseline MAS value of at least one treated indication was available. This OM was analyzed only for participants treated for nasolabial folds.
Measure: Number; unit: percentage of participants
Arm/Group | RADIESSE® (+) Lidocaine: Nasolabial Folds
Number analyzed (Participants) | 202
percentage of participants
  Week 4 | 87.6
  Week 24/28 (Depending Upon Touch-up) | 78.2
  Week 48/52 (Depending Upon Touch-up) | 41.6
  Week 72/76 (Depending Upon Touch-up) | 23.3

6. Secondary Outcome: Responder Rate for Marionette Lines Based on the Blinded Rater's Evaluation on the MMLS at Week 4 (Prior to Optional Touch-up), at Week 24/28, at Week 48/52, and at Week 72/76 (Depending on Touch-up)
Description: The MMLS was to be used to assess the severity of marionette lines. The assessment was performed separately for the left and the right marionette line by the blinded rater and the treating investigator (at baseline only prior to SMD injection) by live rating. MMLS was a 5 point scale ranging from: 0 (no lines), 1 (mild lines), 2 (moderate lines), 3 (severe lines), 4 (very severe lines). Responders rate was defined as percentage of participants who achieved improvement of >=1 point in both marionette lines (left and right) from Day 1 pre-injection to Week 4, Week 24/28, Week 48/52, and Week 72/76 (depending on touch-up). As planned, the cumulative data was collected for Week 24 or 28, Week 48 or 52, and Week 72 or 76 based on the touch-up.
Time Frame: At Week 4 (prior to optional touch-up); and at Weeks 24, 48 and 72 (for participants with no touch-up) or at Weeks 28, 52 and 76 (for participants with touch-up)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | RADIESSE® (+) Lidocaine: Marionette Lines
Number analyzed (Participants) | 194
percentage of participants
  Week 4 | 86.6
  Week 24/28 (Depending Upon Touch-up) | 71.6
  Week 48/52 (Depending Upon Touch-up) | 35.6
  Week 72/76 (Depending Upon Touch-up) | 16.0

7. Secondary Outcome: Responder Rate for Cheek Fullness Based on the Blinded Rater's Evaluation on the MUCFS at Week 4 (Prior to Optional Touch-up), at Week 24/28, at Week 48/52, and at Week 72/76 (Depending on Touch-up)
Description: The MUCFS was used to assess the severity of volume loss of upper cheeks. The assessment was performed separately for the left and the right cheek by the blinded rater and the treating investigator (at baseline only prior to SMD injection) by live rating. MUCFS was based on 5 point scale ranging from: 0 (full upper cheek), 1 (mildly sunken upper cheek), 2 (moderately sunken upper cheek), 3 (severely sunken upper cheek), 4 (very severely sunken upper cheek). Responders rate was defined as percentage of participants who achieved improvement of >=1 point in both cheeks (left and right) from Day 1 pre-injection to Week 4, Week 24/28, Week 48/52, and Week 72/76 (depending on touch-up). As planned, the cumulative data was collected for Week 24 or 28, Week 48 or 52, and Week 72 or 76 based on the touch-up.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | RADIESSE® (+) Lidocaine: Cheek Volume Loss
Number analyzed (Participants) | 188
percentage of participants
  Week 4 | 84.6
  Week 24/28 (Depending Upon Touch-up) | 72.9
  Week 48/52 (Depending Upon Touch-up) | 51.6
  Week 72/76 (Depending Upon Touch-up) | 30.9

8. Secondary Outcome: Number of Participants Based on Treating Investigator's Evaluation of the Global Aesthetic Improvement on the iGAIS at Week 4 (Prior to Optional Touch-up), Week 12/16, Week 24/28, Week 48/52, and Week 72/76 (Depending on Touch-up Performed)
Description: The Investigator's Global Aesthetic Improvement Scale (iGAIS) was used to assess aesthetic improvement in the participants by the treating investigator by live rating using baseline photographs for comparison. The treating investigator was asked: 'Based on your clinical experience, what is your overall impression of change of the participant's aesthetic result due to treatment, compared to the condition before the first treatment (baseline)? Please check the one option that best fits your overall impression of change based on your comparison of the baseline visit photographs.' Rating was based on 7 point rating scale ranging from: +3 (very much improved), +2 (much improved), +1 (improved), 0 (no change), -1 (worse), -2 (much worse), -3 (very much worse). As planned, the cumulative data was collected at Week 4 (prior to optional touch-up), Week 12 or 16, Week 24 or 28, Week 48 or 52, and Week 72 or 76 based on the touch-up.
Time Frame: At Week 4 (prior to optional touch-up); at Weeks 12, 24, 48 and 72 (for participants with no touch-up) or at Weeks 16, 28, 52 and 76 (for participants with touch-up)
Population: The FAS was the subset of all participants who were exposed to the SMD at least once and for whom a baseline and a post-baseline MAS value of at least one treated indication was available. This OM was analyzed in all participants and by the subpopulations of each indication. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure and "number analyzed" were participants who were evaluable for the outcome measure at given time points.
Measure: Count of Participants; unit: Participants
Arm/Group | RADIESSE® (+) Lidocaine: Nasolabial Folds | RADIESSE® (+) Lidocaine: Marionette Lines | RADIESSE® (+) Lidocaine: Cheek Volume Loss | RADIESSE® (+) Lidocaine: All Participants
Number analyzed (Participants) | 201 | 193 | 187 | 205
Participants
  Week 4: Very Much Improved | 24 | 23 | 24 | 26
  Week 4: Much Improved | 106 | 102 | 100 | 107
  Week 4: Improved | 67 | 65 | 60 | 68
  Week 4: No Change | 4 | 3 | 3 | 4
  Week 4: Worse | 0 | 0 | 0 | 0
  Week 4: Much Worse | 0 | 0 | 0 | 0
  Week 4: Very Much Worse | 0 | 0 | 0 | 0
  Week 12/16 (Depending Upon Touch-up): number analyzed (Participants) | 197 | 189 | 183 | 201
  Week 12/16 (Depending Upon Touch-up): Very Much Improved | 32 | 30 | 30 | 32
  Week 12/16 (Depending Upon Touch-up): Much Improved | 115 | 113 | 108 | 118
  Week 12/16 (Depending Upon Touch-up): Improved | 43 | 39 | 40 | 44
  Week 12/16 (Depending Upon Touch-up): No Change | 7 | 7 | 5 | 7
  Week 12/16 (Depending Upon Touch-up): Worse | 0 | 0 | 0 | 0
  Week 12/16 (Depending Upon Touch-up): Much Worse | 0 | 0 | 0 | 0
  Week 12/16 (Depending Upon Touch-up): Very Much Worse | 0 | 0 | 0 | 0
  Week 24/28 (Depending Upon Touch-up): number analyzed (Participants) | 192 | 185 | 178 | 196
  Week 24/28 (Depending Upon Touch-up): Very Much Improved | 6 | 4 | 6 | 6
  Week 24/28 (Depending Upon Touch-up): Much Improved | 86 | 87 | 85 | 89
  Week 24/28 (Depending Upon Touch-up): Improved | 76 | 70 | 68 | 77
  Week 24/28 (Depending Upon Touch-up): No Change | 24 | 24 | 19 | 24
  Week 24/28 (Depending Upon Touch-up): Worse | 0 | 0 | 0 | 0
  Week 24/28 (Depending Upon Touch-up): Much Worse | 0 | 0 | 0 | 0
  Week 24/28 (Depending Upon Touch-up): Very Much Worse | 0 | 0 | 0 | 0
  Week 48/52 (Depending Upon Touch-up): number analyzed (Participants) | 179 | 173 | 166 | 183
  Week 48/52 (Depending Upon Touch-up): Very Much Improved | 1 | 0 | 1 | 1
  Week 48/52 (Depending Upon Touch-up): Much Improved | 13 | 12 | 13 | 13
  Week 48/52 (Depending Upon Touch-up): Improved | 106 | 105 | 100 | 109
  Week 48/52 (Depending Upon Touch-up): No Change | 58 | 55 | 51 | 59
  Week 48/52 (Depending Upon Touch-up): Worse | 1 | 1 | 1 | 1
  Week 48/52 (Depending Upon Touch-up): Much Worse | 0 | 0 | 0 | 0
  Week 48/52 (Depending Upon Touch-up): Very Much Worse | 0 | 0 | 0 | 0
  Week 72/76 (Depending Upon Touch-up): number analyzed (Participants) | 159 | 153 | 148 | 162
  Week 72/76 (Depending Upon Touch-up): Very Much Improved | 0 | 0 | 0 | 0
  Week 72/76 (Depending Upon Touch-up): Much Improved | 6 | 6 | 6 | 6
  Week 72/76 (Depending Upon Touch-up): Improved | 64 | 62 | 61 | 65
  Week 72/76 (Depending Upon Touch-up): No Change | 88 | 84 | 80 | 90
  Week 72/76 (Depending Upon Touch-up): Worse | 1 | 1 | 1 | 1
  Week 72/76 (Depending Upon Touch-up): Much Worse | 0 | 0 | 0 | 0
  Week 72/76 (Depending Upon Touch-up): Very Much Worse | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Based on Participant's Evaluation of the Global Aesthetic Improvement on the sGAIS at Week 4 (Prior to Optional Touch-up), Week 12/16, Week 24/28, Week 48/52, and Week 72/76 (Depending on Touch-up Performed)
Description: The Subject's Global Aesthetic Improvement Scale (sGAIS) was used to assess aesthetic improvement in the participants by the participant by live rating using baseline photographs for comparison. The participant was asked: 'What is your overall impression of change of your aesthetic result due to treatment, compared to the condition before the injection? Please tick the one option that best fits your overall impression of change based on your comparison of the baseline visit photographs.' Rating based on 7 point rating scale ranging from: +3 (very much improved), +2 (much improved), +1 (improved), 0 (no change), -1 (worse), -2 (much worse), -3 (very much worse). As planned, the cumulative data was collected at Week 4 (prior to optional touch-up), Week 12 or 16, Week 24 or 28, Week 48 or 52, and Week 72 or 76 based on the touch-up.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- RADIESSE® (+) Lidocaine: Nasolabial Folds: Participants received SMD (RADIESSE® (+) Lidocaine) on Day 1 with volume and using injection techniques based on investigator's judgement, skin conditions, safety and participant's expectations, and the extent of the volume loss/deficit for treatment of nasolabial folds. An optional touch-up was performed at Week 4 (Visit 2) in the indications that were treated on Day 1, to obtain an optimal aesthetic outcome, as appropriate.
Arm/Group | RADIESSE® (+) Lidocaine: Nasolabial Folds | RADIESSE® (+) Lidocaine: Marionette Lines | RADIESSE® (+) Lidocaine: Cheek Volume Loss | RADIESSE® (+) Lidocaine: All Participants
Number analyzed (Participants) | 201 | 193 | 187 | 205
Participants
  Week 4: Very Much Improved | 9 | 7 | 9 | 9
  Week 4: Much Improved | 71 | 70 | 71 | 75
  Week 4: Improved | 102 | 98 | 89 | 102
  Week 4: No Change | 18 | 17 | 17 | 18
  Week 4: Worse | 0 | 0 | 0 | 0
  Week 4: Much Worse | 0 | 0 | 0 | 0
  Week 4: Very Much Worse | 1 | 1 | 1 | 1
  Week 12/16 (Depending Upon Touch-up): number analyzed (Participants) | 197 | 189 | 183 | 201
  Week 12/16 (Depending Upon Touch-up): Very Much Improved | 20 | 19 | 20 | 20
  Week 12/16 (Depending Upon Touch-up): Much Improved | 84 | 80 | 80 | 87
  Week 12/16 (Depending Upon Touch-up): Improved | 80 | 78 | 73 | 81
  Week 12/16 (Depending Upon Touch-up): No Change | 11 | 10 | 8 | 11
  Week 12/16 (Depending Upon Touch-up): Worse | 0 | 0 | 0 | 0
  Week 12/16 (Depending Upon Touch-up): Much Worse | 1 | 1 | 1 | 1
  Week 12/16 (Depending Upon Touch-up): Very Much Worse | 1 | 1 | 1 | 1
  Week 24/28 (Depending Upon Touch-up): number analyzed (Participants) | 192 | 185 | 178 | 196
  Week 24/28 (Depending Upon Touch-up): Very Much Improved | 8 | 8 | 7 | 8
  Week 24/28 (Depending Upon Touch-up): Much Improved | 61 | 59 | 57 | 63
  Week 24/28 (Depending Upon Touch-up): Improved | 90 | 87 | 86 | 92
  Week 24/28 (Depending Upon Touch-up): No Change | 27 | 26 | 22 | 27
  Week 24/28 (Depending Upon Touch-up): Worse | 5 | 4 | 5 | 5
  Week 24/28 (Depending Upon Touch-up): Much Worse | 1 | 1 | 1 | 1
  Week 24/28 (Depending Upon Touch-up): Very Much Worse | 0 | 0 | 0 | 0
  Week 48/52 (Depending Upon Touch-up): number analyzed (Participants) | 179 | 173 | 166 | 183
  Week 48/52 (Depending Upon Touch-up): Very Much Improved | 0 | 0 | 0 | 0
  Week 48/52 (Depending Upon Touch-up): Much Improved | 26 | 24 | 23 | 26
  Week 48/52 (Depending Upon Touch-up): Improved | 87 | 84 | 82 | 89
  Week 48/52 (Depending Upon Touch-up): No Change | 47 | 46 | 43 | 49
  Week 48/52 (Depending Upon Touch-up): Worse | 16 | 16 | 15 | 16
  Week 48/52 (Depending Upon Touch-up): Much Worse | 1 | 1 | 1 | 1
  Week 48/52 (Depending Upon Touch-up): Very Much Worse | 2 | 2 | 2 | 2
  Week 72/76 (Depending Upon Touch-up): number analyzed (Participants) | 158 | 152 | 147 | 161
  Week 72/76 (Depending Upon Touch-up): Very Much Improved | 1 | 1 | 1 | 1
  Week 72/76 (Depending Upon Touch-up): Much Improved | 20 | 21 | 20 | 21
  Week 72/76 (Depending Upon Touch-up): Improved | 63 | 60 | 57 | 63
  Week 72/76 (Depending Upon Touch-up): No Change | 61 | 57 | 56 | 63
  Week 72/76 (Depending Upon Touch-up): Worse | 11 | 11 | 11 | 11
  Week 72/76 (Depending Upon Touch-up): Much Worse | 2 | 2 | 2 | 2
  Week 72/76 (Depending Upon Touch-up): Very Much Worse | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 72 (for participants with no touch-up) or Week 76 (for participants with touch-up)
Description: The investigator asked the participant for AEs systematically at each visit. As planned, the cumulative data was collected for Week 72 or 76 based on the touch-up.
Arm/Group | RADIESSE® (+) Lidocaine: Nasolabial Folds | RADIESSE® (+) Lidocaine: Marionette Lines | RADIESSE® (+) Lidocaine: Cheek Volume Loss | RADIESSE® (+) Lidocaine: All Participants
All-Cause Mortality (participants affected / at risk) | 0/203 | 0/195 | 0/189 | 0/207
Serious Adverse Events (participants affected / at risk) | 5/203 | 5/195 | 4/189 | 5/207
Other Adverse Events (participants affected / at risk) | 139/203 | 133/195 | 129/189 | 142/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RADIESSE® (+) Lidocaine: Nasolabial Folds (N=203) | RADIESSE® (+) Lidocaine: Marionette Lines (N=195) | RADIESSE® (+) Lidocaine: Cheek Volume Loss (N=189) | RADIESSE® (+) Lidocaine: All Participants (N=207)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1 — Investigator assessed serious adverse event as not related to study treatment.
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 1 — Investigator assessed serious adverse event as not related to study treatment.
Diverticulitis (Infections and infestations) | 1 | 1 | 1 | 1 — Investigator assessed serious adverse event as not related to study treatment.
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 — Investigator assessed serious adverse event as not related to study treatment.
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 — Investigator assessed serious adverse event as not related to study treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RADIESSE® (+) Lidocaine: Nasolabial Folds (N=203) | RADIESSE® (+) Lidocaine: Marionette Lines (N=195) | RADIESSE® (+) Lidocaine: Cheek Volume Loss (N=189) | RADIESSE® (+) Lidocaine: All Participants (N=207)
Injection site haematoma (General disorders) | 79 | 75 | 75 | 81
Injection site swelling (General disorders) | 42 | 39 | 39 | 42
Injection site pain (General disorders) | 13 | 12 | 13 | 13
Injection site nodule (General disorders) | 9 | 9 | 9 | 9
Injection site erythema (General disorders) | 4 | 4 | 4 | 4
Injection site pruritus (General disorders) | 2 | 1 | 2 | 2
Nasopharyngitis (Infections and infestations) | 40 | 38 | 38 | 41
Gastroenteritis (Infections and infestations) | 9 | 9 | 9 | 9
Bronchitis (Infections and infestations) | 7 | 7 | 6 | 7
Sinusitis (Infections and infestations) | 5 | 5 | 5 | 5
Herpes simplex (Infections and infestations) | 2 | 2 | 2 | 2
Pneumonia (Infections and infestations) | 2 | 2 | 2 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 3 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 5 | 5
Headache (Nervous system disorders) | 2 | 2 | 2 | 2
Hypertension (Vascular disorders) | 2 | 2 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03650387/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT03650387/SAP_001.pdf